CLINICAL TRIAL: NCT01706614
Title: Biochemical and Genetic Markers in Liver Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Karolin Hoeh, Study Investigator, University Hospital Heidelberg
Other Study IDs: S-565/2011
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Biochemical and Genetic Markers in Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Investigation of biochemical and genetic markers in liver disease that might have an influence on the course of the disease

ELIGIBILITY:
Inclusion Criteria:

* suffering from liver disease
* age of 18 years or older
* agreement to participate in study

Exclusion Criteria:

* younger than 18 years
* no consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with liver disease seen at department of Gastroenterology, University Hospital Heidelberg
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-04

CONTACTS AND LOCATIONS:
Overall Officials: Karolin J Hoeh, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany